CLINICAL TRIAL: NCT04951609
Title: A Short-term Exploratory Study to Evaluate Safety, Tolerability and Pharmacokinetics of Seltorexant as Adjunctive Therapy to Antidepressants in Adolescents With Major Depressive Disorder Who Have an Inadequate Response to SSRI Monotherapy and Psychotherapy
Brief Title: A Study of Seltorexant as Adjunctive Therapy to Antidepressants in Adolescents With Major Depressive Disorder Who Have an Inadequate Response to Selective Serotonin Reuptake Inhibitor (SSRI) and Psychotherapy
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Following discussion on pediatric strategy with HAs, it was determined that we have sufficient data to inform next steps for the seltorexant pediatric program.
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR109041; 2021-000567-77 (EudraCT Number); 42847922MDD1016 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2021-06-30; First posted 2021-07-07 (Actual); Last update posted 2025-04-27 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — seltorexant

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Seltorexant (Experimental): Participants will receive weight based dose of Seltorexant orally once daily from Day 1 to Day 42 (until the end of Week 6). Participants will continue baseline selective serotonin reuptake inhibitor (SSRI) antidepressant (Fluoxetine or escitalopram) orally once daily.
  Interventions: Drug: Seltorexant
- Placebo (Placebo Comparator): Participants will receive matching placebo tablets to seltorexant orally once daily from Day 1 to Day 42 (until the end of Week 6).
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Seltorexant — Participants will receive a single oral dose of seltorexant.
  Other Names: JNJ-42827922
  Arms: Seltorexant
Drug: Placebo — Participants will receive matching placebo orally.
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the safety and tolerability of Seltorexant as adjunctive therapy to an antidepressant in adolescents with major depressive disorder (MDD) in the short-term compared with placebo.

DETAILED DESCRIPTION:
The prevalence of major depression is approximately 4 percentage (%) to 8% in adolescents, with the highest incidence of MDD in child onset depression occurring during mid- to late adolescence (that is, 14 to 18 years of age). Seltorexant (JNJ-42847922) is a potent and selective antagonist of the human orexin-2 receptor (OX2R) that is being developed for the treatment of adjunctive treatment of MDD with insomnia symptoms (MDDIS).The study will be conducted in 3 phases: a screening phase (up to 30 days prior to first dose administration), a double-blind (DB) treatment phase (6 weeks), and a follow-up phase (up to 2 weeks including a telephone consult and on-site follow-up visit. The total study duration for each participant will be up to 12 weeks. Efficacy, safety, pharmacokinetics, and biomarkers will be assessed at specified time points during this study. The hypothesis for this study is that the safety, tolerability, and pharmacokinetics in the adolescent MDD population. There is no formal statistical hypothesis testing due to the exploratory and descriptive nature of this study.

ELIGIBILITY:
Inclusion Criteria:

* Has inadequate response to trial of at least 1, but no more than 2 antidepressant treatments during the current major depressive episode including their current antidepressant fluoxetine or escitalopram (SSRI). Inadequate response is determined as less than (<) 50 percentage (%) symptom reduction after adequate antidepressant treatment for at least 6 weeks at or above the minimum therapeutic dose prior to screening
* Has had access to adequate psychotherapy in the current depressive episode (based on investigator judgement/local guidance) prior to randomization
* Must have Children's Depression Rating Scale-Revised (CDRS-R) total score greater than or equal to (>=) 48 at screening and >=40 at the baseline visit
* Participants weighing between fifth and ninety-fifth percentile for age and sex. Obese participants greater than ninety-fifth percentile and underweight participants below fifth percentile may participate following medical clearance, as long as their baseline weight is >=30 kilograms (kg)
* A female participant of childbearing potential must have a negative urine pregnancy test at screening and baseline

Exclusion Criteria:

* Has a history of liver or renal insufficiency, significant cardiac (example, congenital heart disease, cardiomyopathy, or tachyarrhythmias), vascular, pulmonary, gastrointestinal, endocrine (including uncontrolled hyperthyroidism), neurologic (including seizure disorder), hematologic, rheumatologic, psychiatric, or metabolic disturbances. Stable medical conditions are allowed
* Has current the diagnostic and statistical manual of mental disorders, fifth edition (DSM-5) diagnosis of conduct disorder, intellectual disability, autism spectrum disorder, borderline personality disorder, somatoform disorders, or fibromyalgia. A prior history of one or more of these disorders is allowed as long as the disorder(s) are currently stable and major depressive disorder (MDD) is not secondary to the original diagnosis. Has a current or prior DSM-5 diagnosis of a psychotic disorder, or bipolar disorder
* Has a significant primary sleep disorder (example, obstructive sleep apnea, parasomnias) at screening but participants with insomnia or hypersomnia disorders are allowed
* At significant risk of committing suicide based on history or according to the investigator's experience, or based on active suicidal ideation, intent or plan, item 4 or 5 of the Columbia-Suicide Severity Rating Scale (C-SSRS) within the past 3 months or a history of suicidal behavior within the last 6 months
* Has known allergies, hypersensitivity, or intolerance to seltorexant or its excipients

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2021-09-02 (Actual); Primary Completion 2024-04-08 (Actual); Study Completion 2024-04-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Treatment Emergent Adverse Events (TEAEs) | Up to 12 weeks
  An adverse event is any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. TEAEs are adverse events with onset during the double-blind treatment phase or that are a consequence of a preexisting condition that has worsened since baseline.
Number of Participants with Adverse Event of Special Interest (AESIs) | Up to 12 weeks
  Number of participants with AESIs will be reported. AEs are considered to be of special interest in this study: a) Cataplexy (sudden, transient episode of muscle weakness accompanied by conscious awareness); b) Sleep paralysis (the experience of not being able to move, react, or speak when falling asleep/awakening); c) Complex, sleep-related behaviors/parasomnias such as confusional arousals, somnambulism (sleep walking), sleep terrors, bruxism (teeth grinding), sleep sex, sleep-related eating disorder, and catathrenia (REM-associated end-inspiratory apnea/breath holding); d) Any new suicidal behavior or suicidal ideation.
Pediatric Adverse Event Rating Scale (PAERS) | Up to 12 weeks
  The PAERS is a patient-rated scale designed to assess adverse events occurring in pediatric participants treated with psychotropic medication in clinical studies. Individual PAERS (patient-reported version) will rate symptoms and severity of symptoms. This scale has a total of 48 items. There is no overall score and individual item will be rated on a scale of 0 to 4 in which 0 indicates 'not present' and 4 indicates 'very bothersome/an extreme problem'.
Number of Participants with Abnormalities in Clinical Laboratory Values | Up to 6 weeks
  Number of participants with abnormalities in clinical laboratory values (hematology, serum chemistry and urinalysis) will be reported.
Number of Participants with Abnormalities in Electrocardiogram (ECG) | up to 6 weeks
  Number of participants with abnormalities in ECG will be reported.
Number of Participants with Abnormalities in Vital Signs | Up to 12 weeks
  Number of participants with abnormalities in vital sign(blood pressure and pulse/heart rate) will be reported.
Number of Participants with Abnormalities in Physical Examination | Up to 6 weeks
  Number of participants with abnormalities in physical examination including weight will be reported.
Suicidality Assessment Using the Columbia Suicide Severity Rating Scale (C-SSRS) Score | Up to 12 weeks
  Suicidality assessment using the C-SSRS will be reported. C-SSRS is a clinician rated assessment of suicidal behavior and/ or intent. Scale consists of 28 items in 4 sections: suicide behavior, actual attempts, suicidal ideation, and intensity of ideation. Suicidal ideation consists of 5 yes/no items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, active suicidal ideation with specific plan and intent. Worsening of suicidal ideation will be an increase in severity of suicidal ideation from baseline.
Withdrawal Symptoms Assessment Using the Physician Withdrawal Checklist (PWC-20) | 2 weeks
  Withdrawal symptoms assessment using the PWC-20 will be reported. The PWC-20 is a simple and accurate method used to assess potential withdrawal symptoms following cessation of treatment. The PWC-20 is a reliable and sensitive instrument for the assessment of discontinuation symptoms. Each individual item score ranges from 0 (not present) to 3 (severe), where higher scores = more affected condition.
Number of Participants with Menstrual Cycle Tracking | Up to 6 weeks
  Number of participants with menstrual cycle tracking will be reported. Menstrual cycles will be tracked during the study in female adolescents or participants who have at least one menses using a participant diary and participant's verbal report.

SECONDARY OUTCOMES:
Change from Baseline to Week 6/End of Treatment (EOT) in the Children's Depression Rating Scale (CDRS) Total Score | Baseline up to 6 weeks
  Change from baseline to week 6/EOT in the CDRS total score will be reported. The CDRS-R is a validated 17-item, clinician-rated instrument that measures the severity of a participant's depressive symptoms. The CDRS-R total score is the sum of the responses to 17 questions. Each question is graded on a 5- or 7-point scale. The highest possible score is 113 (the most severe measure of depression), and the lowest is 17 (not suffering from depression).
Change from Baseline to Week 6 in Montgomery Asberg Depression Rating Scale (MADRS) Score | Baseline up to 6 weeks
  Change from baseline in MADRS score will be reported. The 10-item MADRS is a clinician-administered scale designed to measure depression severity and detects changes due to antidepressant treatment. The test consists of 10 items, each of which is scored from 0 (item not present or normal) to 6 (severe or continuous presence of the symptoms), for a total score of 60. Higher score represents a more severe condition.
Change from Baseline in Clinical Global Impression- severity (CGI-S) Score Over Time | Baseline up to 6 weeks
  Change from baseline over time in the CGI-S score will be reported. The CGI-S provides an overall clinician-determined summary measure of the severity of the participant's illness. The CGI-S evaluates the severity of psychopathology on a scale of 1 to 7. Considering total clinical experience with the depression population, a participant is assessed on severity of illness at the time of rating according to: 1=normal (not at all ill); 2=borderline ill; 3=mildly ill; 4=moderately ill; 5=markedly ill; 6=severely ill; 7=among the most extremely ill participants.
Change from Baseline to Week 6/EOT on Subjective Sleep Assessment (Patient Reported Outcome Measurement Information System-Pediatric-Sleep Disturbance [PROMIS-Pediatric-SD] [Short Form 8a]) | Baseline up to 6 weeks
  Change from baseline to week 6/EOT on subjective sleep assessment (PROMIS-Pediatric-SD [short form 8a]) will be reported. The PROMIS-SD is used to assess self-reported perceptions of sleep quality, sleep depth and restoration associated with sleep. The full PROMIS-SD includes 27 items with each item based on a 7-day recall period and assessed on a 5 level Likert-type scale. The 8-item short form will be used in this study, in which responses are scored 1 to 5 for each item. A higher score on 5 of the 8 items reflects a worse outcome, whereas a higher score on 3 items reflects an improved outcome; therefore, the directionality of the 8 item scores is first synchronized prior to calculation of the total raw score. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. Higher overall score indicates more sleep disturbance.
Change from Baseline to Week 6/EOT on Objective Sleep Assessment Actigraphy | Baseline up to 6 weeks
  Change from baseline to week 6/EOT on objective sleep assessment actigraphy will be reported. The primary purpose of actigraphy in this study is to have an objective measure of sleep parameters prior to treatment to complement the Consensus Sleep Diary (CSD) as well as other sleep-related PROs.
Cognitive Performance on a Neurocognitive Battery at Baseline and Week 6/EOT | Baseline, Week 6
  The cogstate computerized cognitive battery is a validated set of assessments which will be performed to assess verbal learning and memory and evaluate cognitive function. The battery will provide assessment of multiple cognitive domains, including attention, visual learning and memory, and executive function. All measures in the cognitive battery have been validated against traditional neuropsychological tests and are sensitive to the effects of various drugs on cognitive performance, including alcohol and benzodiazepines. The participants completed Cogstate computerized cognitive battery has been used for cognitive assessment in several child and adolescent research trials including attention deficit hyperactivity disorder, and demonstrates good reliability and validity in child and adolescent populations. The ISLT has also been used in adolescent trials, demonstrating sensitivity, reliability and validity.
Change in Subjective Sleep Related Impairment (PROMIS-Pediatric- Sleep-Related Impairment [SRI]) | Up to 6 weeks
  Change in subjective sleep related impairment (PROMIS-Pediatric-SRI) will be reported. The PROMIS_SRI is used to assess self reported daytime sleepiness and impact on functioning. . The full PROMIS-SD includes 27 items with each item based on a 7-day recall period and assessed on a 5 level Likert-type scale. The 8-item short form will be used in this study, in which responses are scored 1 to 5 for each item. A higher score on 5 of the 8 items reflects a worse outcome, whereas a higher score on 3 items reflects an improved outcome; therefore, the directionality of the 8 item scores is first synchronized prior to calculation of the total raw score. To find the total raw score for a short form with all questions answered, sum the values of the response to each question. Higher overall score indicates more sleep disturbance.
Plasma Concentration of Seltorexant | Up to 6 weeks
  Plasma concentration of seltorexant will be reported using a validated, specific, and sensitive liquid chromatography/mass spectrometry/mass spectrometry (LC-MS/MS) method.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (23):
- United States (12):
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - Advanced Research Center Inc, Anaheim, California
  - University of California at San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - Sarkis Clinical Trials, Gainesville, Florida
  - APG Research LLC, Orlando, Florida
  - Baber Research Group, Naperville, Illinois
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - CincyScience, West Chester, Ohio
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
- Italy (3):
  - G.Gaslini Institute, Genova
  - Ospedale Pediatrico Bambin Gesù, Roma
  - Universita Cattolica del Sacro Cuore - Fondazione Policlinico Universitario 'A. Gemelli', Roma
- Spain (6):
  - Hosp. Sant Joan de Deu, Esplugues de Llobregat
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Clinica Univ. de Navarra Madrid, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Majadahonda
  - Corporacio Sanitari Parc Tauli, Sabadell
- United Kingdom (2):
  - South London and Maudsley NHS Foundation Trust of The Maudsley Hospital, London
  - Warneford Hospital, NIHR Clinical Research Facility, Oxford

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency